CLINICAL TRIAL: NCT06925412
Title: Sponge Application of MMC Versus Suntenon Injection in Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hazem Elbadry Mohammed Mohammed, Lecturer of Ophthalmology, Department of Ophthalmology, Faculty of Medicine, Benha University, Egypt, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ophth._27/2024Med.Research
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-01

CONDITIONS: Trabeculectomy; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMC sponge application (Experimental)
  Interventions: Procedure: MMC sponge application
- Sub-Tenon MMC injection (Experimental)
  Interventions: Procedure: Sub-tenon MMC injection

INTERVENTIONS:
Procedure: MMC sponge application — Three micro swabs soaked in 0.03% MMC were subconjunctivally applied, followed by the creation of a fornix-based conjunctival flap. Subsequently, the standard trabeculectomy procedure was initiated without additional irrigation of the MMC application site
  Arms: MMC sponge application
Procedure: Sub-tenon MMC injection — MMC was administered via a sub-tenon injection. A 30-gauge needle was inserted into the conjunctiva and carefully advanced laterally along Tenon's capsule. A cannula was employed to minimize the excessive spread of MMC over the anticipated conjunctival incision site. After MMC delivery, a fornix-based conjunctival peritomy was performed, and both groups proceeded to undergo standard trabeculectomy
  Arms: Sub-Tenon MMC injection

SUMMARY:
Glaucoma is a leading cause of irreversible blindness worldwide, with intraocular pressure (IOP) reduction being the primary therapeutic goal. Trabeculectomy, augmented with mitomycin C (MMC), remains the gold standard surgical intervention but is limited by postoperative fibrosis. MMC delivery methods, including sponge application and sub-Tenon injection, vary in drug distribution and may influence surgical outcomes. This study aimed to compare the efficacy and safety of trabeculectomy using sponge-applied MMC versus sub-Tenon MMC injection, focusing on IOP reduction, bleb morphology, and postoperative medication requirements.

In this retrospective, randomized controlled trial, 50 patients with primary or secondary glaucoma were assigned to trabeculectomy with either MMC sponge application (Group A, n=25) or sub-Tenon MMC injection (Group B, n=25). All surgeries were performed by the same surgeon using standardized techniques. Patients were followed for one year, with primary outcomes including IOP reduction and secondary outcomes encompassing bleb morphology (Indiana Bleb Appearance Grading Scale), bleb integrity (Seidel test), and postoperative glaucoma medication use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* diagnosed with primary open-angle glaucoma (POAG) or secondary glaucoma,
* uncontrolled IOP (IOP > 21 mmHg) despite maximally tolerated medical therapy,
* progressive visual field deterioration,
* or intolerance to anti-glaucoma medications.

Exclusion Criteria:

* age under 18 years,
* absence of light perception,
* previous incisional glaucoma surgery,
* need for combined ocular procedures,
* intraoperative use of 5-fluorouracil (5-FU),
* or follow-up duration of less than one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) reduction | One year

SECONDARY OUTCOMES:
Bleb morphology (Indiana Bleb Appearance Grading Scale) | One year
Bleb integrity (Seidel test) | One year
Postoperative glaucoma medication use | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Ebsar Eye Center, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdelhafeez SME, Mohammed Mohammed HE, Tharwat E, Ibrahim MM, Tawfik AMR, Elgohary RMA, Alabshihy MSI, Sakr AM, Ebrahim AM, Mohammed AR, Yusef NM, Saliem EA, Elsayed SSE, Elsayed Saad EM. Sponge Application of Mitomycin C vs Sub-Tenon Injection in Trabeculectomy: A Randomized Controlled Trial. J Curr Glaucoma Pract. 2025 Oct-Dec;19(4):199-207. doi: 10.5005/jp-journals-10078-1500. Epub 2025 Dec 15. PMID 41523175